CLINICAL TRIAL: NCT02362204
Title: Development and Feasibility of a Lung Cancer Nurse Model During Early Treatment: a Phase II Study
Brief Title: Lung Cancer Nurse Model: a Phase II Study
Acronym: LCN-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Freiburg (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Dr Manuela Eicher, Dean of research School of Health Sciences Fribourg-HEdS-FR, University of Freiburg
Other Study IDs: UniversityFreiburg
Record Dates: First submitted 2015-02-07; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: therapeutic education and psychological support — Intervention consists of alternate face-to-face consultations (anticipated duration: 60-90 minutes) and telephone consultations (anticipated duration: 15-30 minutes). All interventions will include: i) a focused assessment of physical and psychological symptoms, ii) information about lung cancer (disease) and its treatment, iii) a review of disease-related and treatment-related side effects and strategies to manage these symptoms, and iv) printed listing and review of available support resources.

SUMMARY:
Lung cancer patients experience significant physical symptoms, psychological distress and have many supportive care needs that impact on quality of life. Implementing the role of a Lung Cancer Nurse (LCN) is a response to meet the needs of patients and caregivers.

Primary aim is to assess the feasibility of a LCN intervention and feasibility to collect longitudinal patient self-assessment questionnaires at the Thoracic Cancer Centre of the University Hospital of Lausanne.

Secondary aims are: i) to describe self-reported changes in self-efficacy, symptoms and unmet supportive care needs across three time points during the first line therapy and ii) to explore professional acceptability of the new LCN model evaluating the perceptions of barriers and facilitators of the model by the LCN and the other multidisciplinary members of the comprehensive lung cancer care team.

An exact single-stage (no interim analysis) design will be applied to determine feasibility for further studies to be undertaken. Secondary outcomes will be analyzed descriptively at each data collection (Baseline, Time1, Time2) time point and professional acceptability will be explored by focus groups with selected members of the interdisciplinary team.

DETAILED DESCRIPTION:
To develop adequate self-care strategies, patients with lung cancer and their families are in need of emotional, informational and behavioural supportive care. Supportive care in cancer can reduce symptom burden and improve patients and their families self-management skills. As lung cancer incidence continues to rise, and increased attention is given to early diagnosis, research on early involvement of lung cancer nurse (LCN) in care, the feasibility and impact on patient outcomes is needed.

Primary aim is to assess the feasibility of a LCN intervention and feasibility to collect longitudinal (Baseline, Time1, Time2) patient self-assessment questionnaires at the Thoracic Cancer Centre of the University Hospital of Lausanne.

Secondary aims are: i) to describe self-reported changes in self-efficacy, symptoms and unmet supportive care needs across three time points during the first line therapy and ii) to explore professional acceptability of the new LCN model evaluating the perceptions of barriers and facilitators of the model by the LCN and the other multidisciplinary members of the comprehensive lung cancer care team.

An exact single-stage (no interim analysis) design will be applied to determine feasibility for further studies to be undertaken. Lung cancer patients with planned systemic therapy with or without radiotherapy will be recruited at the thoracic cancer center in a Swiss University Hospital. The LCN model of care consists of two face-to-face consultations alternating with two telephone consultations during systemic therapy. LCN consultations will comprise focused assessment of physical and psychological symptoms, information (printed and oral) about disease and its treatment, therapeutic education concerning strategies to manage physical and psychosocial symptoms and review of available support resources. Participants will be invited to complete the validated patient reported Lung Cancer Symptom Scale, Supportive Care Needs Screening Tool 9 and Self-Efficacy Scale for Lung Cancer. Study data will be collected at baseline (day 1 of systemic therapy), time 1 (week 3 of systemic therapy) and time 2 (week 11 of systemic therapy). Participants will be categorized as adherent if they complete all their scheduled LCN consultations and questionnaires. For a 5% probability of accepting a poor feasibility (alpha) and a 20% probability of rejecting an acceptable feasibility (beta) we then need to enroll 71 patients. Feasibility will be considered as acceptable for further studies if at least 36 patients will be compliant. Secondary outcomes will be analyzed descriptively for each variable (self-efficacy, symptoms and supportive care needs) across each time point. At the end of quantitative data collection, a focus group will be conducted to explore acceptability of the new role among health professionals working with the LCN in order to identify perceived barriers and facilitators for collaborative work with the new role.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed lung cancer (NSCLC or SCLC)
* Patients capable of speaking and writing in French
* Patients undergoing programmed a systemic treatment (with or without radiotherapy treatment)
* Estimated life expectancy more than 6-months
* Signing the written informed consent document

Exclusion Criteria:

* Patients diagnosed with lung cancer receiving only surgery treatment or only a radiotherapy treatment
* Patients not physically or emotionally capable of participating in the trial as determined by their oncologist (existing mental illness or severe physical disability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients newly diagnosed receiving systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 11 weeks
  For a 5% probability of accepting a poor feasibility and a 20% probability of rejecting an acceptable feasibility we need to enroll 71 patients. Feasibility will be considered as acceptable for further studies if at least 36 patients reach the end of the study completing their scheduled Lung Cancer Nurse consultations and patients completed the three questionnaire at each data collect time (baseline, time 1 and time 2)

SECONDARY OUTCOMES:
Lung cancer symptoms | Baseline-Week 3- Week 11
  Symptoms will be measured by the Lung Cancer Symptom Scale .This inventory consists of 9 items relating to appetite, fatigue, cough, dyspnea, hemoptysis, and pain related to lung malignancies and three summary items on symptom distress, interference with activity level, and global health-related quality of life. Each item is scored on a visual scale 0-100 (0=no symptom; 100 symptom as bad as can be).
Unmet Supportive Care Need | Baseline-Week 3- Week 11
  Unmet Supportive Care Needs will be measured by the the Supportive Care Needs Survey Screening Tool 9 (SCNS ST 9). The 9 items of the scale fall into five analytically derived factor domains: i) psychological, ii) health system and information, iii) physical and daily living, iv) patient care and support, and v) sexuality. Each item is rated on a 5-point Likert-type scale (not applicable=1; satisfied=2; low need=3; moderate need=4; High need=5).
Self-efficacy | Baseline-Week 3- Week 11
  Self-efficacy will be measured by the Self-Efficacy Scale for lung cancer. This scale is composed by 16 items regarding patients' perceived ability to manage a variety of symptoms on a scale of 10 (not at all certain) to 100 (completely certain). The instrument includes three subscale concerning: i) self-efficacy for managing pain, ii) self-efficacy for managing other symptoms, and iii) self-efficacy for functions.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Eicher, Dr, Study Director — University of Freiburg
Locations (1):
- University Hospital of Lausanne, Lausanne, Switzerland